CLINICAL TRIAL: NCT05276856
Title: Rate of Recovery of Secondary Hypothyroidism in Patients With Pituitary Disorders.
Brief Title: Recovery Rate in Secondary Hypothyroidism
Status: Recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: RR in secondary hypothyroidism
Record Dates: First submitted 2022-02-28; First posted 2022-03-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Secondary Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Levothyroxine — Step 1:
  * Reduce the dose of T4 therapy by 50% and recheck serum T4 after 2 weeks.
  * If serum T4 is normal, go to step 2.
  * If serum T4 drops to below normal then resume full T4 replacement (these patients will be considered as having withdrawal failure).
  Step 2:
  * Discontinue T4 therapy altogether and recheck serum TSH and T4 after 2 weeks.
  * If serum T4 is normal, go to step 3.
  * If serum T4 drops to below normal then resume full T4 replacement (these patients will be considered as having withdrawal failure).
  Step 3:
  * Recheck serum TSH and T4 after 8 weeks.
  * If serum TSH and T4 levels are normal, these patients will be regarded as having successful T4 withdrawal.
  * If T4 drops to below normal then resume full T4 replacement (these patients will be considered as having withdrawal failure).

SUMMARY:
The aim of this project is to assess the rate of recovery of secondary hypothyroidism in patients with pituitary disorders.

DETAILED DESCRIPTION:
The study will be conducted in three stages.

Stage 1 ( Patient identification and enrollment)

We will generate a list of all SHT patients from the HNP database and all patients will be contacted by the principal investigator (or their designate) regarding the study. Those patients who agree to participate in the study will be given a written consent form. We aim to enrol approximately 90 -100 patients for the study. Laboratory samples for serum TSH and T4 levels will be collected to confirm that all patients are adequately replaced for SHT. Those patients who are not adequately replaced and have low T4 will be excluded from the study.

Stage 2 (T4 withdrawal protocol)

Stepwise T4 replacement therapy will be initiated as follows.

Step 1:

* Reduce the dose of T4 therapy by 50% and recheck serum T4 after 2 weeks.
* If serum T4 is normal, go to step 2.
* If serum T4 drops to below normal then resume full T4 replacement (these patients will be considered as having withdrawal failure).

The rationale for testing serum T4 after 2 weeks is that the half life of T4 is up to 7 days and early testing will potentially give false results. Furthermore, serum T3 is not a reliable test in patients taking T4 therapy and will not be requested 6.

Step 2:

* Discontinue T4 therapy altogether and recheck serum TSH and T4 after 2 weeks.
* If serum T4 is normal, go to step 3.
* If serum T4 drops to below normal then resume full T4 replacement (these patients will be considered as having withdrawal failure).

Step 3:

* Recheck serum TSH and T4 after 8 weeks.
* If serum TSH and T4 levels are normal, these patients will be regarded as having successful T4 withdrawal.
* If T4 drops to below normal then resume full T4 replacement (these patients will be considered as having withdrawal failure).

Stage 3 (Analysis)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of secondary hypothyroidism who are currently taking T4 replacement therapy

Exclusion Criteria:

* uncontrolled cardiovascular disease
* uncontrolled congestive heart failure
* uncontrolled mental health disorder
* not adequately replaced and have low T4 level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with pituitary disorders in the province of Nova Scotia are routinely enrolled in a computerized registry called the Halifax Neuropituitary (HNP) database. The database currently contains information on approximately 1800 patients. All pituitary hormonal dysfunctions are routinely identified in the HNP database. For this study, we will identify all patients with confirmed diagnosis of SHT who are currently taking T4 replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving euthyroid status | 12 weeks
  Percentage of patients able to maintain normal TSH/T4 without thyroxine replacment

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Canada

REFERENCES:
- [Background] Al-Dahmani K, Mohammad S, Imran F, Theriault C, Doucette S, Zwicker D, Yip CE, Clarke DB, Imran SA. Sellar Masses: An Epidemiological Study. Can J Neurol Sci. 2016 Mar;43(2):291-7. doi: 10.1017/cjn.2015.301. Epub 2015 Nov 2. PMID 26522017
- [Background] Munro V, Tugwell B, Doucette S, Clarke DB, Lacroix A, Imran SA. Recovery of adrenal function after chronic secondary adrenal insufficiency in patients with hypopituitarism. Clin Endocrinol (Oxf). 2016 Aug;85(2):216-22. doi: 10.1111/cen.13048. Epub 2016 Mar 21. PMID 26928716
- [Background] Hudec M, Grigerova M, Walsh CH. Secondary hypothyroidism in hereditary hemochromatosis: recovery after iron depletion. Thyroid. 2008 Feb;18(2):255-7. doi: 10.1089/thy.2007.0140. PMID 18205549
- [Background] Hwang JY, Aum DJ, Chicoine MR, Dacey RG Jr, Osbun JW, Rich KM, Zipfel GJ, Klatt-Cromwell CN, McJunkin JL, Pipkorn P, Schneider JS, Silverstein JM, Kim AH. Axis-specific analysis and predictors of endocrine recovery and deficits for non-functioning pituitary adenomas undergoing endoscopic transsphenoidal surgery. Pituitary. 2020 Aug;23(4):389-399. doi: 10.1007/s11102-020-01045-z. PMID 32388803
- [Background] Zhang R, Wang Z, Gao L, Guo X, Feng C, Deng K, Lian W, Yao Y, Feng M, Bao X, Wang R, Xing B. Clinical Characteristics and Postoperative Recovery of Hypopituitarism in Patients with Nonfunctional Pituitary Adenoma. World Neurosurg. 2019 Jun;126:e1183-e1189. doi: 10.1016/j.wneu.2019.03.062. Epub 2019 Mar 14. PMID 30880207
- [Background] Livingston M, Birch K, Guy M, Kane J, Heald AH. No role for tri-iodothyronine (T3) testing in the assessment of levothyroxine (T4) over-replacement in hypothyroid patients. Br J Biomed Sci. 2015;72(4):160-3. doi: 10.1080/09674845.2015.11665746. PMID 26738396